CLINICAL TRIAL: NCT04668222
Title: Based on the Theory of "Body Constitution of Chinese Medicine" and "Combination of Prescription and Syndrome" to Improve COVID-19 Susceptible Body Constitution of Residents in Hong Kong
Brief Title: Changing Susceptible Body Constitution for COVID-19 Prevention by Chinese Medicine in Hong Kong Residents
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor FENG Yibin, Professor Feng Yibin, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UW20-480
Record Dates: First submitted 2020-11-30; First posted 2020-12-16 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: COVID19; Herbal Medicine
Keywords: COVID19 Prevention; Chinese Medicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: According to the assessment of "Self-test for classification and judgment of body constitution by TCM theory", participants with the body constitution of "deficiency of Qi and Yin" or "deficiency of Qi and Yin" will be included into this study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Deficiency of Qi and Yang (QYang-group) (Experimental): Participants will receive Yu-Ping-Feng and Xiang-Sha-Liu-Jun formula (Chinese Medicine Formula)
  Interventions: Drug: Yu-Ping-Feng formula; Drug: Xiang-Sha-Liu-Jun formula
- Placebo control of invigorating Qi and Yang (PQYang-group) (Placebo Comparator): The placebo is made of 5% Yu-Ping-Feng and Xiang-Sha-Liu-Jun formula (Chinese Medicine Formula)
  Interventions: Drug: Placebo for "Deficiency of Qi and Yang"
- Deficiency of Qi and Yin (QYin-group) (Experimental): Participants will receive Yu-Ping-Feng and Liu-Wei-Di-Huang formula (Chinese Medicine Formula)
  Interventions: Drug: Yu-Ping-Feng formula; Drug: Liu-Wei-Di-Huang formula
- Placebo control of invigorating Qi and Yin (PQYin-group) (Placebo Comparator): The placebo is made of 5% Yu-Ping-Feng and Liu-Wei-Di-Huang formula (Chinese Medicine Formula)
  Interventions: Drug: Placebo for "Deficiency of Qi and Yin"

INTERVENTIONS:
Drug: Yu-Ping-Feng formula — Yu-Ping-Feng formula produced by PuraPharm International (H.K) Ltd is a registered Chinese medicine formula by Chinese Medicine Council of Hong Kong (registration number: HKC-08255). The intake dosage is 5g twice daily.
  Arms: Deficiency of Qi and Yang (QYang-group); Deficiency of Qi and Yin (QYin-group)
Drug: Xiang-Sha-Liu-Jun formula — Xiang-Sha-Liu-Jun formula produced by PuraPharm International (H.K) Ltd is a registered Chinese medicine formula by Chinese Medicine Council of Hong Kong (registration number: HKC-08252). The intake dosage is 5g twice daily.
  Arms: Deficiency of Qi and Yang (QYang-group)
Drug: Liu-Wei-Di-Huang formula — Liu-Wei-Di-Huang formula produced by PuraPharm International (H.K) Ltd is a registered Chinese medicine formula by Chinese Medicine Council of Hong Kong (registration number: HKC-08273). The intake dosage is 5g twice daily.
  Arms: Deficiency of Qi and Yin (QYin-group)
Drug: Placebo for "Deficiency of Qi and Yang" — Placebo for the group of "deficiency of Qi and Yang" is composed of 5% Yu-Ping-Feng formula+Xiang-Sha-Liu-Jun formula
  Arms: Placebo control of invigorating Qi and Yang (PQYang-group)
Drug: Placebo for "Deficiency of Qi and Yin" — Placebo for the group of "deficiency of Qi and Yin" is composed of 5% Yu-Ping-Feng formula+Liu-Wei-Di-Huang formula
  Arms: Placebo control of invigorating Qi and Yin (PQYin-group)

SUMMARY:
Chinese medicine has been used for thousands of years in the treatment of epidemic diseases. Through the long-term struggle with the epidemic, Investigators have accumulated and explored a lot of prevention and control experience. According to recent reports, Chinese medicine plays an important role in the treatment of COVID-19. For example. Therefore, it is of great clinical significance to further develop the prevention of COVID-19 by Chinese medicine. According to the 《Diagnosis and treatment of COVID-19》published by National Health Committee and the experience of professional TCM physician, although the disease is generally susceptible, individuals with the body constitution of "deficiency of Qi and Yang" and "deficiency of Qi and Yin" are more prefer to suffer from COVID-19. Therefore, "Invigorating Qi and Yang, invigorating qi and Yin" can be regarded as the primary strategy of preventing COVID-19. Therefore, "Invigorating Qi and Yang, invigorating qi and Yin" can be regarded as the primary strategy of preventing COVID-19 in Chinese medicine. After a series of questionnaire surveys and blood sample collection, investigators can estimate subjects with body constitution is more likely to infect COVID-19.

DETAILED DESCRIPTION:
In December 2019, COVID-19 has been outbreaks in a series regions of China and abroad. Its pathogen was initially identified as a new coronavirus with single strand positive RNA. COVID-19 is considered to be a coronavirus associated with severe acute respiratory syndrome (SARS) and Middle East respiratory syndrome (MERS), which can affect the lower respiratory tract and manifest as pneumonia. On January 31, 2020, the World Health Organization (WHO) officially announced that COVID-19 has become a "public health emergency of international concern" Although most provinces in China have inhibited the spread of COVID-19 after taking protective measures, the number of patients worldwide is still on the rise. According to WHO and recent reports, On 1st Sept, 2020, the total number of clinically confirmed cases in the world is 25327098, and the current total number in China is 90402. China has incorporated COVID-19 into the class B infectious diseases in the law on the prevention and control of infectious diseases. Notably, it adopted the prevention and control of class A infectious diseases. It is worth noting that residents of Hong Kong have also been seriously infected with COVID-19. According to the latest report released by the Department of Health in Hong Kong, the total number of patients with COVID-19 had risen to 4823 on Sept 1st, 2020. Therefore, it is very urgent to find effective control methods.

According to the theory of Chinese medicine, COVID-19 belongs to the category of "epidemic toxin". TCM has been used for thousands of years in the treatment of epidemic diseases. Through the long-term struggle with the epidemic, investigators have accumulated a lot of experience for the pathogenesis, transmission, prevention and control of the epidemic. In mainland China, TCM plays an important role in the treatment of COVID-19. The recent retrospective analysis of 52 cases by Zhang Boli's research group showed that 34 cases in the treatment group of integrated TCM and Western medicine were superior to 18 cases in the simple western medicine group in terms of various bio-indexes, including clinical symptoms disappearance, the time of body temperature recovery, the average length of stay in hospital, the score of TCM Syndrome Scale, the rate of CT image improvement, the rate of clinical cure, and the conversion from common type to severe type. According to a case study of 799 people in Hunan Provincial Administration of traditional Chinese medicine, the average length of stay in hospital of integrated traditional Chinese and Western medicine treatment is 2 days shorter than that of Western medicine treatment alone, and the number of patients with obvious improvement of symptoms accounts for 64% of the total number of observation. For the modern measures of epidemic prevention, it includes three approaches: cutting off pathogens, controlling transmission routes, and reducing susceptible populations. However, so far, the preventive measures of Chinese medicine for COVID-19 has not been included in the medical system of Hong Kong, although it is widely authorized and promoted in mainland China. Therefore, it is of great clinical significance to further develop the prevention of COVID-19 by Chinese medicine for reducing susceptible populations. The National Health Committee and the State Administration of TCM organized relevant experts to establish COVID-19 standardized diagnosis and treatment program. The updated diagnosis and treatment program describes the relationship between the dialectical classification of Chinese medicine and the stage of Western medicine. The pathogenesis of TCM can be summarized as "dampness, heat, toxin, blood stasis, deficiency". According to the statement of Tong Xiaolin, COVID-19 belongs to "cold dampness epidemic", which is caused by cold dampness epidemic virus. The disease is mainly caused by the deficiency of either yin or Yang. According to a report on the clinical epidemiology of COVID-19 published by Lancet, the median susceptible population of COVID-19 is 49 years old (interquartile range is 41-58 years old), which means the majority of patients are middle-aged and elderly. The body constitution of this kind of patients is mainly divided into " Deficiency of Qi and Yang " and "Deficiency of Qi and Yin". However, so far, the prevention of treatment of COVID-19 with TCM has not been included in the medical system of Hong Kong, although TCM therapy is widely authorized and promoted in mainland China. Therefore, It may be beneficial to provide TCM preventive measures to COVID-19 in Hong Kong. By using "Self-test for classification and judgment of body constitution by TCM theory" issued by Professor Wang Qi, a honorary Professor of School of Chinese medicine, the University of Hong Kong, investigators can identify the subjects with "Deficiency of Qi and Yang " or "Deficiency of Qi and Yin". According to the above-mentioned pathogenesis characteristics of COVID-19 in the prevention stage, "Invigorating Qi and Yang, invigorating Qi and Yin" may be conducted by TCM treatment. The changes of body constitution will be measured by questionnaires before and after TCM intervention, including Self-test for classification and judgment of body constitution by TCM theory, Questionnaire of TCM symptom, and Fatigue scale.

In order to scientifically evaluate the preventive effect of TCM on COVID-19, it is very important to reveal the changes of COVID-19 related biochemical indexes before and after the intervention of TCM. According to the discussion on 《Diagnosis and treatment of COVID-19》issued by the National Health Commission, the following changes in biochemical indicators are closely related to the occurrence of COVID-19. Firstly, the decrease of leukocytes, lymphocytes, and bone marrow cells (including granulocytes, erythrocytes, and megakaryocytes) in blood routine examination; the increase of troponin and ESR. Secondly, the reduction of macrophages-related immune cells, such as monocyte. Thirdly, the increased index of liver function and cardiac function, including AST, ALT, and LDH. Fourthly, inflammation related factors, including IL-6 and C-reactive protein. Therefore, the analysis of the relationship model of TCM syndrome and molecular biological profiles can further provide a novel preventive mode for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above, regardless of gender;
2. For COVID-19 susceptible individuals, according to the criteria of "Self-test for classification and judgment of body constitution by TCM theory", subjects with deficiency of Qi with either Yin or Yang will meet the inclusion criteria;
3. No previous allergy to traditional Chinese medicine;
4. Be able to understand Chinese questionnaire;
5. Willing to participate in the study.

Exclusion Criteria:

1. Syndrome types are not related to "deficiency of Qi and Yang" and "deficiency of Qi and Yin";
2. Suspected or confirmed COVID-19 patients;
3. Fever, body temperature > 37°C with cough and other respiratory symptoms;
4. Those who have visited the epidemic area and have not completed isolation for 14 days after returning to Hong Kong

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Potential COVID-19 susceptible body constitutions will be measured by the scale of "Self-test for classification and judgment of body constitution by traditional Chinese medicine (TCM) theory" | 1 month
  At the beginning of the clinical trial, the classification of body constitution will be determined by scale of "Self-test for classification and judgment of body constitution by Traditional Chinese Medicine (TCM) theory", in which 8 kinds of body constitutions are involved, including the potential COVID-19 susceptible body constitution "deficiency of Qi with either Yang and Yin". There are 9 types of body constitution and 7 choices for each body constitution. The minimun and maximum score for each body constitution is 7 and 35, respectively. The total score of this scale is 315. Higer score in a specific item stands for the stonger correlation with a specific body constitution.
Changes of TCM-based syndromes will be measured by the "Questionnaire of TCM symptom" | 1 month
  The scale of "Questionnaire of Traditional Chinese Medicine (TCM) symptom" will be used to measure the changes of TCM specific symtom before and after the treatment, such as the changes of "Irritable motion" and " insomnia". The scale of "Questionnaire of TCM symptom" consists of 20 items and each item has 4 choices. The minimun and maximum score for each body is 1 and 4, respectively. The total score of this scale is 80. Higer score in a specific item represents the stonger correlation with a specific TCM symptom
Potential changes of fatigue status will be measured by Fatigue Scale | 1 month
  The fatigue scale is a 13-item scale of fatigue status. Items are scored on a 0 to 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the fatigue, all items are summed to create a single fatigue score ranging from 0 to 52. Higer score stands for a stonger correlation with fatigue.

SECONDARY OUTCOMES:
Complete Blood Count will be measured by Automated Cell Counter | 1 month
  According to the "Diagnosis and treatment of new coronavirus pneumonia (7th Edition)" published by National Health Commission of China, the investigators will measure the potential COVID19-fluctuated Complete Blood Count (red blood cells, white blood cells, and platelets), before and after the treatment.
Liver function biomarkers in blood will be measured by Automatic Blood Biochemistry Analyzer | 1 month
  In terms of the "Diagnosis and treatment of new coronavirus pneumonia (7th Edition)", the investigators will further test the potential COVID19-fluctuated liver biomarkers by Automatic Blood Biochemistry Analyzer, including aspartate aminotransferase (AST) and alanine aminotransferase (ALT), before and after the treatment.
Heart function biomarkers in blood will be measured by Automatic Blood Biochemistry | 1 month
  According to the "Diagnosis and treatment of new coronavirus pneumonia (7th Edition)", the investigators will further test the potential COVID19-fluctuated heart biomarkers by Automatic Blood Biochemistry Analyzer, including lactate dehydrogenase (LDH), troponin I,before and after the treatment.
Inflammatory biomarker in blood will be measured by Automatic Blood Biochemistry | 1 month
  In accordance with the "Diagnosis and treatment of new coronavirus pneumonia (7th Edition)", the investigators will measure the inflammatory biomarker IL-6 by Automatic Blood Biochemistry, which is widely involved in the pathogenesis of several inflammations.
The changes of quantification of blood CD4 and CD8 populations will be measured by flow cytometric analyzer | 1 month
  For futher analyzing the potential COVID19-fluctuated immuno-markers, the investigators will measure the population of CD4, CD8, and CD4/CD8 ratio in the blood by flow cytometric analyzers. The biomarkers of CD4 and CD8 will be used to stain the blood cells followed by the detection of its populations.
Kidney function biomarker, blood urea (dL/L), will be measured by Automatic Blood Biochemistry | 1 month
  According to the "Diagnosis and treatment of new coronavirus pneumonia (7th Edition)", the investigators will further test the potential COVID19-fluctuated kidney biomarkers by Automatic Blood Biochemistry Analyzer, including blood urea before and after the treatment.
Kidney function biomarker, creatinine in blood (μmol/L), will be measured by Automatic Blood Biochemistry | 1 month
  According to the "Diagnosis and treatment of new coronavirus pneumonia (7th Edition)", the investigators will further test the potential COVID19-fluctuated kidney biomarkers by Automatic Blood Biochemistry Analyzer, including blood creatinine before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yibin Feng, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sohrabi C, Alsafi Z, O'Neill N, Khan M, Kerwan A, Al-Jabir A, Iosifidis C, Agha R. World Health Organization declares global emergency: A review of the 2019 novel coronavirus (COVID-19). Int J Surg. 2020 Apr;76:71-76. doi: 10.1016/j.ijsu.2020.02.034. Epub 2020 Feb 26. PMID 32112977
- [Result] Mahase E. Coronavirus covid-19 has killed more people than SARS and MERS combined, despite lower case fatality rate. BMJ. 2020 Feb 18;368:m641. doi: 10.1136/bmj.m641. No abstract available. PMID 32071063
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT04668222/Prot_001.pdf
  • Informed Consent Form (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT04668222/ICF_000.pdf